CLINICAL TRIAL: NCT07016737
Title: Immunochemotherapy ± Salvage Chemoradiation for Local Recurrence of Esophageal Squamous Cell Carcinoma After Definitive Chemoradiotherapy (ESO-Nanjing12)
Brief Title: Immunochemotherapy ± Salvage Chemoradiation for Local Recurrence of Esophageal Squamous Cell Carcinoma After Definitive Chemoradiotherapy
Acronym: ESO-Nanjing12
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ye jinjun (Other)
Responsible Party: Sponsor-Investigator, Ye jinjun, Chief Physician, M.D., Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-008-01; 2024-008-01 (Registry Identifier: ESO-Nanjing12)
Record Dates: First submitted 2025-05-15; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Esophageal squamous cell carcinoma; Local recurrence at the primary tumor site; Programmed cell death protein 1; Salvage Chemoradiotherapy; Immunochemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Carboplatin; Omeprazole; Dexamethasone; Loperamide; atropine sulfate-diphenoxylate hydrochloride drug combination; High-Energy Shock Waves; Gastroscopy

STUDY DESIGN:
Intervention Model Description: The study will focus on those who have attained a complete response (CR) subsequent to definitive chemoradiotherapy or radiotherapy and have a histologically proven in-field recurrence, with no distant metastases. These patients will receive treatment with a PD-1 inhibitor (sintilimab or camrelizumab 200mg, d1, q3w) combined with monotherapy chemotherapy (paclitaxel 175mg/m2 or docetaxel 75mg/m2 or irinotecan 270mg/m2, d1, q3w) for 4 cycles, followed by a 2-year maintenance treatment with PD-1 inhibitors. During this period, patients diagnosed with esophageal wall thickening and identified as having progressive disease (PD) have the option to undergo salvage radiotherapy (45-50.4 Gy/25-28/F/5-5.5 weeks) in conjunction with a dual-agent chemotherapy (paclitaxel 50 mg/m2, d1 + carboplatin AUC 2, d1, qw) for 5 cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): This is a prospective clinical study designed to enroll 79 patients. The study will focus on those who have attained a complete response (CR) subsequent to definitive chemoradiotherapy or radiotherapy and have a histologically proven in-field recurrence, with no distant metastases. These patients will receive treatment with a PD-1 inhibitor (sintilimab or camrelizumab 200mg, d1, q3w) combined with monotherapy chemotherapy (paclitaxel 175mg/m2 or docetaxel 75mg/m2 or irinotecan 270mg/m2, d1, q3w) for 4 cycles, followed by a 2-year maintenance treatment with PD-1 inhibitors. During this period, patients diagnosed with esophageal wall thickening and identified as having progressive disease (PD) have the option to undergo salvage radiotherapy (45-50.4 Gy/25-28/F/5-5.5 weeks) in conjunction with a dual-agent chemotherapy (paclitaxel 50 mg/m2, d1 + carboplatin AUC 2, d1, qw) for 5 cycles.
  Interventions: Drug: Sintilimab Combined With Docetaxel Monotherapy

INTERVENTIONS:
Drug: Sintilimab Combined With Docetaxel Monotherapy — 79 patients will receive treatment with a PD-1 inhibitor (sintilimab or camrelizumab 200mg, d1, q3w) combined with monotherapy chemotherapy (paclitaxel 175mg/m2 or docetaxel 75mg/m2 or irinotecan 270mg/m2, d1, q3w) for 4 cycles, followed by a 2-year maintenance treatment with PD-1 inhibitors. During this period, patients diagnosed with esophageal wall thickening and identified as having progressive disease (PD) have the option to undergo salvage radiotherapy (45-50.4 Gy/25-28/F/5-5.5 weeks) in conjunction with a dual-agent chemotherapy (paclitaxel 50 mg/m2, d1 + carboplatin AUC 2, d1, qw) for 5 cycles.
  Other Names: Sintilimab Combined With Paclitaxel Monotherapy; Sintilimab Combined With Irinotecan Monotherapy; Camrelizumab Combined With Docetaxel Monotherapy; Camrelizumab Combined With Paclitaxel Monotherapy; Camrelizumab Combined With Irinotecan Monotherapy; Paclitaxel Combined With Carboplatin; salvage radiotherapy; Omeprazole; Dexamethasone; Smectite Powder; Loperamide Hydrochloride Capsules; Atropine Hydrochloride; Computed Tomography; Positron Emission Tomography - Computed Tomography; Ultrasound; Gastroscopy; Digital Gastrointestinal Radiography

SUMMARY:
The combination of programmed death receptor 1 (PD-1) inhibitors with chemotherapy has been recognized for the treatment of advanced and metastatic esophageal squamous cell carcinoma (ESCC). To the best of our knowledge, there is no published report to date which analyzes the efficacy and safety of this regimen in the treatment of locally primary-recurrent ESCC patients after definitive chemoradiotherapy or radiotherapy only. This is a prospective clinical study designed to enroll 79 patients. The study will focus on those who have attained a complete response (CR) subsequent to definitive chemoradiotherapy or radiotherapy and have a histologically proven in-field recurrence, with no distant metastases. These patients will receive treatment with a PD-1 inhibitor combined with monotherapy chemotherapy for 4 cycles, followed by a 2-year maintenance treatment with PD-1 inhibitors. During this period, patients diagnosed with esophageal wall thickening and identified as having progressive disease (PD) have the option to undergo salvage radiotherapy in conjunction with a dual-agent chemotherapy for 5 cycles. The primary endpoint of is 2-year after recurrence survival (ARS) rate. The secondary endpoints include the progression-free survival (PFS) and safety.

ELIGIBILITY:
Inclusion Criteria:

-1.Age ≥18 years, regardless of gender. 2.Pathologically confirmed local recurrence of esophageal squamous cell carcinoma after definitive chemoradiotherapy.

3.With or without regional lymph node metastasis, but no distant metastasis. 4.Ineligible for surgery or refusal to undergo surgical intervention. 5.Tolerance to chemotherapy, radiotherapy, and immunotherapy. 6.ECOG performance status 0-2. 7.Life expectancy ≥3 months. 8.No severe hematopoietic, cardiac, pulmonary, hepatic, renal dysfunction, or immunodeficiency.

Exclusion Criteria:

* 1. Esophageal perforation or hematemesis. 2.Distant metastasis in patients after definitive chemoradiotherapy. 3.History of drug abuse, chronic alcoholism, or HIV/AIDS. 4.Myocardial infarction within ≤6 months. Patients with myocardial infarction >6 months ago must undergo myocardial thallium scan to confirm absence of myocardial ischemia and obtain cardiologist approval for chemotherapy.

  5.Uncontrolled seizures or psychiatric disorders impairing decision-making capacity.

  6.Severe allergic history or hypersensitivity. 7.Other conditions deemed unsuitable for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
2-year ARS rate | From date of Immunochemotherapy until the date of death from any cause, assessed up to 24 months
  the proportion of patients surviving 2 years from the time of recurrence

SECONDARY OUTCOMES:
progression-free survival (PFS) | From date of Immunochemotherapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  From Initiation of Immunochemotherapy to Disease Progression
safety assessed by adverse events (TEAEs) | Up to 2 years after treatment initiation until new treatment
  All treatment-emergent adverse events (TEAEs) related to the investigational drug were documented and graded according to the CTCAE v5.0 criteria during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Ye jin jiun, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Provincial Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No